CLINICAL TRIAL: NCT01687621
Title: Omphalitis Community Based Algorithm Validation Study
Acronym: OCAVS
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Julie M Herlihy, Assistant Professor, Boston University
Other Study IDs: OCAVS
Record Dates: First submitted 2012-09-07; First posted 2012-09-19 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Omphalitis
Keywords: Omphalitis; Neonate; Zambia; Neonatal mortality; Umbilical cord infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates, 1 to 10 days old: Neonates between day 1-10 of life presenting to hospitals and community health centers in Southern Province, Zambia, with no prior diagnosis of omphalitis, whose guardian, aged 15 and above, is willing to allow their newborn to participate in the study.
  Interventions: Procedure: Diagnostic Algorithm for Community Based Worker for Omphalitis

INTERVENTIONS:
Procedure: Diagnostic Algorithm for Community Based Worker for Omphalitis — After obtaining guardian informed written consent, newborns aged 1-10 days presenting to the health facility for routine or sick visits would undergo 2 independent, parallel evaluations; first, by a ZamCAT Field Monitor (community level worker from our existing study) and the second by a Zambian medical doctor (gold standard). A US board of pediatrics-certified pediatrician will perform a third independent assessment of a photo of the cord remotely. Using the on-site clinician as the gold standard, the community-based algorithm and the photo assessment will be tested for concordance and the sensitivity and specificity of the algorithm will be generated. Likewise, the remote pictorial assessment will be compared to the gold standard to determine reliability of diagnosis from photographs alone.

SUMMARY:
The objective of this study is to develop and test a simple community-based diagnostic algorithm for omphalitis in sub-Saharan Africa. To date, there has been no validated community-based algorithms developed and tested in the sub-Saharan context where the manifestations of omphalitis presentation may vary and diagnosis could be potentially more challenging in infants with darker skin color. Given the current attention to cord care at the global and national policy level, validated community-based algorithms will be needed to allow primary health workers to identify cord infections and reduce associated morbidity.

After obtaining guardian informed consent, newborns aged 1-10 days presenting to the health facility for routine or sick visits will undergo two independent, parallel evaluations; first, by a community level worker and second, by a Zambian medical doctor (gold standard). A third independent assessment of a photo of the cord will be performed remotely by a board-certified pediatrician. Using the on-site clinician as the gold standard, the community-based algorithm and the photo assessment will be tested for concordance and the sensitivity and specificity of the algorithm will be generated. Likewise, the remote pictorial assessment will be compared to the gold standard to determine reliability of diagnosis from photographs alone.

ELIGIBILITY:
Inclusion Criteria:

* Neonate between day 1-10 of life presenting to Livingstone and Mazabuka district hospitals and community health centers in Southern Province, Zambia
* No prior diagnosis of omphalitis
* Guardian willing to allow their newborn to participate in the study
* Guardian aged 15 and above

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonate between day 1-10 of life presenting to Livingstone and Mazabuka district hospitals and community health centers in Southern Province, Zambia
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Validity of the omphalitis algorithm | 10 months
  The primary outcome of the study is a measure of validity (concordance) of the the omphalitis algorithm generated by inter-observer kappa statistics to evaluate diagnostic concordance between the field monitors and the gold standard cord health expert on specific algorithmic questions. Questions that demonstrate high concordance will be selected for inclusion in the final algorithm. Sensitivity and specificity of the final algorithm will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Herlihy, MD MPH, Principal Investigator — Boston University
Locations (1):
- Hospitals & Community Health Centers, Livingstone, Southern Province, Zambia

REFERENCES:
- See also: Zambia Chlorhexidine Application Trial — http://www.bu.edu/cghd/our-work/projects/zambia-chlorhexidrine-application-trial-zamcat/